CLINICAL TRIAL: NCT00439140
Title: Safety and Efficacy Study of Botulinum Toxin Type A for the Treatment of Neurogenic Overactive Bladder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In agreement with FDA the study was terminated based on data available.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-082
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- botulinum toxin Type A 200U (Experimental): Botulinum toxin Type A 200U injection into the detrusor on Day 1 followed by a repeat botulinum toxin Type A 200U injection after a minimum of 12 weeks (if applicable).
  Interventions: Biological: botulinum toxin Type A
- botulinum toxin Type A 300U (Experimental): Botulinum toxin Type A 300U injection into the detrusor on Day 1 followed by a repeat botulinum toxin Type A 300U injection after a minimum of 12 weeks (if applicable).
  Interventions: Biological: botulinum toxin Type A
- Placebo/botulinum toxin Type A 200U (Other): Placebo (Normal Saline) injection into the detrusor on Day 1 followed by a botulinum toxin Type A 200U injection after a minimum of 12 weeks (if applicable).
  Interventions: Biological: botulinum toxin Type A; Drug: Normal Saline (Placebo)
- Placebo/botulinum toxin Type A 300U (Other): Placebo (Normal Saline) injection into the detrusor on Day 1 followed by a botulinum toxin Type A 300U injection (200U after discontinuation of 300U) after a minimum of 12 weeks (if applicable).
  Interventions: Biological: botulinum toxin Type A; Drug: Normal Saline (Placebo)

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A injection into the detrusor.
  Other Names: BOTOX®; onabotulinumtoxinA
Drug: Normal Saline (Placebo) — Placebo (Normal Saline) injection into the detrusor.
  Arms: Placebo/botulinum toxin Type A 200U; Placebo/botulinum toxin Type A 300U

SUMMARY:
This study will assess the safety and efficacy of botulinum toxin Type A for the treatment of urinary incontinence overactive bladder in patients with a spinal cord injury or multiple sclerosis.

DETAILED DESCRIPTION:
Botulinum toxin Type A 300U has been discontinued from the study after regulatory approval of botulinum toxin Type A 200U. Patients remaining in the study who were allocated to receive botulinum toxin Type A 300U at treatment 2 (and had not yet received it) will receive botulinum toxin Type A 200U instead.

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence as a result of neurogenic overactive bladder due to spinal cord injury or multiple sclerosis
* Inadequate response to anticholinergic medication used to treat overactive bladder.
* Neurological respiratory impairment and abnormal pulmonary function test results

Exclusion Criteria:

* History or evidence of pelvic or urologic abnormality
* Previous or current diagnosis of bladder or prostate cancer
* Symptomatic or untreated urinary tract infection at time of enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Philadelphia, Pennsylvania, United States
- Herston, Queensland, Australia
- Victoria, British Columbia, Canada
- Chennai, India

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Botulinum toxin Type A 300U was discontinued from the study after regulatory approval of botulinum toxin Type A 200U. Patients remaining in the study who were allocated to receive botulinum toxin Type A 300U at treatment 2 (and had not yet received it) received botulinum toxin Type A 200U instead.
Groups:
- Placebo: Placebo (Normal Saline) injection into the detrusor on Day 1. (If applicable after 12 weeks, participants received either botulinum toxin Type A 200U or 300U in Treatment Cycle 2.)
Period: Treatment Cycle 1
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Started | 15 | 14 | 12
Completed | 14 | 10 | 11 (5 patients did not enter Cycle 2. 6 patients received botulinum toxin Type A in Cycle 2.)
Not Completed | 1 | 4 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Personal reasons | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Treatment Cycle 2
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Started | 13 (8 patients from the 200U arm plus 5 patients from the placebo arm in Cycle 1 entered Cycle 2.) | 7 (6 patients from the 300U arm plus 1 patient from the placebo arm in Cycle 1 entered Cycle 2.) | 0 (No patients received placebo in Cycle 2.)
Completed | 11 | 6 | 0
Not Completed | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Botulinum Toxin Type A: Placebo (Normal Saline) injection into the detrusor on Day 1 followed by a botulinum toxin Type A 200U or 300U injection after a minimum of 12 weeks (if applicable).
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo/Botulinum Toxin Type A | Total
Number analyzed (Participants) | 15 | 14 | 12 | 41
Age, Customized [Number; unit: participants]
  < 40 Years | 9 | 8 | 6 | 23
  40-64 Years | 4 | 6 | 6 | 16
  ≥ 65 Years | 2 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 3 | 16
  Male | 8 | 8 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: Spirometry was conducted according to American Thoracic Society standards. A spirometer was used to measure FVC, the maximum amount of air exhaled from the lungs after taking the deepest breath possible, at Baseline and Week 6. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Week 6
Population: Safety Population included all randomized participants who received treatment.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Placebo: Placebo (Normal Saline) injection into the detrusor on Day 1.
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Number analyzed (Participants) | 15 | 14 | 12
Liters
  Baseline | 2.659 (0.5308) | 2.955 (0.7733) | 3.095 (0.6868)
  Change from Baseline at Week 6 | -0.124 (0.2758) | -0.096 (0.2248) | -0.025 (0.2391)

2. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1)
Description: Spirometry was conducted according to American Thoracic Society standards. A spirometer was used to measure FEV1, the maximum amount of air exhaled in one second, at Baseline and Week 6. The highest value at each time-point was recorded. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Week 6
Population: Safety population included all randomized participants who received treatment.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Number analyzed (Participants) | 15 | 14 | 12
Liters
  Baseline | 2.290 (0.5815) | 2.534 (0.7227) | 2.535 (0.7626)
  Change from Baseline at Week 6 | -0.067 (0.2525) | -0.094 (0.2196) | -0.052 (0.1926)

3. Primary Outcome: Change From Baseline in FEV1/FVC Ratio
Description: The FEV1/FVC ratio was calculated by dividing the FEV1 value by the FVC value representing the portion (or ratio) of FVC exhaled in one second. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Week 6
Population: Safety population included all randomized participants who received treatment.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Number analyzed (Participants) | 15 | 14 | 12
Ratio
  Baseline | 0.857 (0.1093) | 0.857 (0.1214) | 0.818 (0.1574)
  Change from Baseline at Week 6 | 0.017 (0.0668) | -0.007 (0.0578) | -0.018 (0.0676)

4. Secondary Outcome: Change From Baseline in the Number of Urinary Incontinence Episodes
Description: The number of urinary incontinence episodes or leakage occurring over the previous 3 days was recorded in the patient bladder diary at Baseline and prior to Week 6. A negative change from Baseline indicated improvement (less incontinence/leakage).
Time Frame: Baseline, Week 6
Population: Participants from the Intent-to-treat population (all randomized participants) using observed data for analysis.
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Number analyzed (Participants) | 15 | 13 | 11
Episodes
  Baseline | 12.5 (9.78) | 13.5 (6.48) | 9.3 (6.59)
  Change from Baseline at Week 6 (n=13,11,11) | -10.2 (7.70) | -9.5 (6.96) | -3.4 (4.57)

5. Secondary Outcome: Change From Baseline in the Maximum (Amplitude) Detrusor Pressure (MDP)
Description: MDP was measured at the first involuntary detrusor contraction using urodynamic testing. A catheter was inserted into the bladder at Baseline and Week 6 and the pressure [measured in centimeters water (cm H20)] was determined as the bladder filled. A negative change from Baseline indicated improvement (less Detrusor pressure).
Time Frame: Baseline, Week 6
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Number analyzed (Participants) | 15 | 14 | 12
cm H2O
  Baseline | 39.1 (30.45) | 42.6 (22.65) | 41.9 (18.91)
  Change from Baseline at Week 6 (n=4,9,9) | -23.3 (28.96) | 0.3 (32.67) | 8.7 (23.91)

6. Secondary Outcome: Change From Baseline in Maximum Cystometric Capacity (MCC)
Description: MCC (the maximum amount of urine the bladder could hold) was measured using urodynamic testing. The amount of urine collected was subtracted from the total volume infused measured as milliliters (mL) of urine. A positive change from Baseline indicated improvement (fuller bladder/ less incontinence).
Time Frame: Baseline, Week 6
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Number analyzed (Participants) | 15 | 14 | 12
mL
  Baseline | 161.4 (80.29) | 216.7 (168.41) | 266.2 (191.41)
  Change from Baseline at Week 6 (n=12,13,11) | 213.2 (135.58) | 60.2 (222.35) | -64.5 (136.98)

7. Other Pre Specified Outcome: Number of Participants With at Least a 15% Decrease From Baseline in FVC
Description: Spirometry was conducted according to American Thoracic Society standards. A spirometer was used to measure FVC, the maximum amount of air exhaled from the lungs after taking the deepest breath possible at Baseline, Weeks 2, 6 and 12.
Time Frame: Baseline, Weeks 2, 6 and 12
Population: Safety population included all randomized participants who received treatment.
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Number analyzed (Participants) | 15 | 14 | 12
Participants
  Week 2 (n=15,14,12) | 0 | 1 | 1
  Week 6 (n=15,14,12) | 2 | 1 | 0
  Week 12 (n=14,12,9) | 0 | 1 | 0

8. Other Pre Specified Outcome: Number of Participants With at Least a 20% Decrease From Baseline in FVC
Description: as for outcome 7
Time Frame: Baseline, Weeks 2, 6 and 12
Population: Safety population included all randomized participants who received treatment.
Measure: Number; unit: Participants
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo
Number analyzed (Participants) | 15 | 14 | 12
Participants
  Week 2 (n=15,14,12) | 0 | 1 | 0
  Week 6 (n=15,14,12) | 1 | 0 | 0
  Week 12 (n=14,12,9) | 0 | 1 | 0

ADVERSE EVENTS:
Description: Serious Adverse Events (SAEs) and Adverse Events (AEs) were reported based on the treatment the participant received. SAEs and AEs reported for participants in the Placebo/Botulinum Toxin Type A arm may have occurred while the participant received placebo in Cycle 1 or botulinum toxin Type A in Cycle 2.
Arm/Group | Botulinum Toxin Type A 200U | Botulinum Toxin Type A 300U | Placebo/Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 4/15 | 6/14 | 1/12
Other Adverse Events (participants affected / at risk) | 12/15 | 12/14 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A 200U (N=15) | Botulinum Toxin Type A 300U (N=14) | Placebo/Botulinum Toxin Type A (N=12)
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 — Event not related to treatment.
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 — Event not related to treatment.
Cellulitis (Infections and infestations) | 1 | 0 | 0
Leptospirosis (Infections and infestations) | 1 | 0 | 0
Typhoid fever (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 — Event not related to treatment.
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 — Event not related to treatment.
Renal function test abnormal (Investigations) | 0 | 1 | 0 — Event not related to treatment.
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 — Event not related to treatment.
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 — Event not related to treatment.
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Botulinum Toxin Type A 200U (N=15) | Botulinum Toxin Type A 300U (N=14) | Placebo/Botulinum Toxin Type A (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Syringomyelia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Thyroid cyst (Endocrine disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 5 | 1
Asthenia (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 9 | 8 | 9
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 — Events not related to treatment.
Influenza (Infections and infestations) | 2 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 — Event not related to treatment.
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 — Event not related to treatment.
Vulvovaginal mycotic infection (Infections and infestations) | 2/7 | 0/6 | 0/3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Leptospirosis (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Typhoid fever (Infections and infestations) | 1 | 0 | 0
Viral rhinitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 — Event not related to treatment.
Septic shock (Infections and infestations) | 0 | 0 | 1 — Event not related to treatment.
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 — Event not related to treatment.
Vaginal infection (Infections and infestations) | 0/7 | 0/6 | 1/3
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Renal function test abnormal (Investigations) | 0 | 1 | 0 — Event not related to treatment.
Residual urine volume (Investigations) | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Pulmonary function test decreased (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 2 — Events not related to treatment.
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1 — Events not related to treatment.
Bladder pain (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 — Event not related to treatment.
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0 | 0 — Event not related to treatment.
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 — Event not related to treatment.
Epididymitis (Reproductive system and breast disorders) | 0/8 | 1/8 | 0/9
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1/7 | 0/6 | 0/3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.